CLINICAL TRIAL: NCT06442774
Title: Digital Tool to Improve Maternal Mental Health: Enhancing Well-being, Early Detection, Diagnosis Support, and Monitoring of Mental Health Problems During the Perinatal Period
Brief Title: MamaConecta: Digital Tool for Maternal Mental Health
Acronym: DDT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: A Thousand Colibris, S.L (Industry)
Collaborators: Hospital Universitari Vall d'Hebron Research Institute (VHIR) (Unknown); Universitat Rovira i Virgili (URV) (Unknown); Hospital del Mar Research Institute (IMIM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ATC/CT001/2023
Record Dates: First submitted 2024-05-14; First posted 2024-06-04 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Pregnancy Related; Mental Health Issue; Postpartum Depression; Postpartum Anxiety; Well-Being, Psychological
Keywords: mental health; pregnancy; mobile application; wellbeing; child neurodevelopment; antenatal depression screening; early detection; postpartum; digital health
MeSH Terms: conditions — Depression, Postpartum; Psychological Well-Being

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will download an app that will randomise them on the intervention or control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Participants of this group will have care as usual from healthcare providers. Participants will have the study variables measured (by questionnaires and monitoring via wearable).
  Interventions: Other: Monitoring via wearable
- Mobile application (Experimental): Participants of this group will have access to the content of the application and will use it regularly from the start of the study until 4 months postpartum. Participants will have the study variables measured (by questionnaires and monitoring via wearable)
  Interventions: Other: Mobile application; Other: Monitoring via wearable

INTERVENTIONS:
Other: Mobile application — The intervention that has been developed is a digital tool of a biopsychosocial nature based on the main cognitive-behavioral strategies: psychoeducation, reflection, self-observation, guided visualizations, mindfulness and progressive muscle relaxation.
  The intervention consists of 3 main areas of work:
  * Programs: Biopsychosocial programs in text and audio format.
  * Community: Forum with directed questions and space to share experiences between mothers.
  * Diary: Space to record mood and emotional record.
  The entire tool works transversally in 4 dimensions: self-care, relationship with perinatal changes, relationship with the baby, social relationship.
  The tool itself includes 3 mental health and well-being screening questionnaires: Whooley Questionnaire and the Edinburgh Postnatal Depression Scale (EPDS).
  Arms: Mobile application
Other: Monitoring via wearable — Participants that own a wearable will connect it to monitor variables related to sleeping patterns, activity and stress (see variables section).

SUMMARY:
The goal of this randomized controlled trial is to validate a digital health tool, Dana app, that enhances well-being and supports mental health monitoring for women during the perinatal period. The primary purpose is to improve maternal well-being, early detection of mental health issues, and aid in the diagnosis and monitoring by healthcare professionals in women transitioning into motherhood. The main questions it aims to answer are:

* Does the app improve overall maternal well-being during the perinatal period?
* Can the app increase the early detection rates of perinatal mental health disorders?
* Can the app be an effective tool to support healthcare professionals to diagnose perinatal mental health problems?
* How effective is the app in improving obstetric outcomes and the psychological and cognitive development of infants?

Researchers will compare the group using the app with a control group not using the digital tool to see if Dana provides significant improvements in maternal and infant health outcomes.

Participants will:

* Use the mobile application from 12-14 weeks of gestation until 24 months postpartum.
* Undergo regular assessments to monitor their emotional state, lifestyle, clinical, and obstetric data.
* Participate in evaluations for their infants' psychological and cognitive development at various stages from birth to two years old.

This trial is conducted at multiple centers, including Hospital Vall d'Hebron, the Sexual and Reproductive Health Care Services (ASSIR) in Tarragona and ASSIR Litoral (Barcelona), Hospital del Mar, following CONSORT standards. The study aligns with the Health and Culture priorities of the Spanish Government's Scientific, Technical, and Innovation Research Plan 2021-2023.

DETAILED DESCRIPTION:
BACKGROUND:

Mental disorders are becoming one of the major health problems in today's society, exacerbated in women who are and will become mothers. Global studies indicate that 80% of women who are going to become mothers experience mood disorders such as stress, fear, loneliness, or guilt during the perinatal period. In 1 out of every 5 cases, these mental disorders worsen and lead to severe mental health issues such as post-traumatic stress disorder, psychosis, suicidal ideation, or postpartum depression. However, 75% of women with perinatal mental disorders are underdiagnosed and do not receive adequate treatment, either due to a lack of detection or support within healthcare systems. This has a consequent impact on the health and well-being of the mother, her family, the child, and ultimately, society. In this context, the company A Thousand Colibris S.L (ATC) has developed digital health software to improve well-being during this period, as well as to detect, assist in the diagnosis, and monitor mental health disorders in mothers from pregnancy up to two years after childbirth.

Consequences of Perinatal Mental Health Disorders:

The consequences of perinatal mental health problems extend beyond the mother, affecting the child, the family, and society as a whole.

1. Maternal health disorders: Perinatal mental health disorders have been identified in women of all cultures, ages, social levels, and races. Although the term postpartum depression is often used to describe disorders that develop after childbirth, a range of disorders can appear during pregnancy and the postpartum period, including anxiety, depression, stress disorders, panic, or postpartum psychosis. If left untreated, these illnesses can have a devastating impact on women and their families, being one of the leading causes of maternal death during pregnancy and the two years following childbirth.
2. Impact on the future health of the child: Without appropriate intervention, these disorders can persist and have negative consequences for both the mother and the baby. The impact of the mother's health on the future health of the baby, on mother-newborn interactions, breastfeeding difficulties, and the mother-child bond is well documented. The failure to detect certain aspects of maternal health can manifest in complications during childbirth or later in the child's development.
3. Impact on family well-being: The mother's mood and symptoms of anxiety and other disorders also have a direct impact on the partner, who may not understand what is happening, feel overwhelmed, and not know how to help.

Digital psychological interventions:

Given the growing ubiquity of the Internet and the widespread use of smartphones, mindfulness-based cognitive-behavioral interventions can also be offered digitally. In this regard, researchers have been successfully adapting decades-old techniques commonly used in cognitive-behavioral therapies to the context of smartphone applications, which have demonstrated efficacy in reducing symptoms of depression, anxiety, stress, insomnia, and even suicidal thoughts. However, the potential of smartphone applications in promoting well-being, and preventing and treating mental health problems in pregnant women, has yet to be fully exploited. Despite the limited number of studies and controlled trials involving health apps for pregnant women, online app stores are flooded with pregnancy apps that have not been tested using rigorous scientific methods. This has sparked an increasing debate among researchers and policymakers regarding the evaluation of quality and certification of health apps that do not meet the needs of patients and doctors, particularly concerning safety and efficacy. Health applications should be evaluated with the same rigor as other types of interventions, such as pharmacotherapy and psychotherapy.

HYPOTHESES:

Hypothesis 1: Dana is a digital tool that improves the well-being of women transitioning into motherhood and increases the early detection of mental health disorders.

Hypothesis 2 (Class IIa Certification): The tool provides monitoring of maternal health and assists in diagnosis for healthcare professionals.

OBJECTIVES:

General:

To validate a digital tool as a solution to (a) improve maternal well-being, mental and physical health during the perinatal period, (b) increase early detection of maternal mental health disorders, and (c) assist in the diagnosis and monitoring of perinatal mental health problems.

Specific:

* Validate the effectiveness of the digital tool in improving well-being at the end of pregnancy (34 weeks gestation), initial postpartum (6 weeks postpartum), and long-term (6, 12, and 24 months postpartum).
* Verify the effectiveness of the digital tool in preventing symptoms of anxiety and depression during the perinatal period (pregnancy and postpartum up to 24 months postpartum).
* In women with symptoms detected in the baseline assessment, analyze the effectiveness of the tool in preventing symptom escalation.
* In women with stabilized mental pathology, analyze the effectiveness of the tool in preventing symptom escalation.
* Verify the effectiveness of the digital tool in improving secondary outcomes related to childbirth: childbirth experience and postpartum-related post-traumatic stress.
* Verify the effectiveness of the digital tool in improving obstetric and neonatal health secondary outcomes.
* Analyze the use of healthcare services and the cost of perinatal mental health.
* Verify the effectiveness of the intervention developed to increase prenatal bonding and postpartum attachment.
* Verify the effectiveness of the intervention developed to improve postpartum secondary outcomes: satisfaction with the maternal role, self-efficacy, stress with the maternal role, and proportion of breastfeeding.
* Analyze the secondary relationship between childbirth experience, post-traumatic stress, and postpartum depression.
* Analyze the data collected by the digital tool and wearables to identify patterns and correlations that may be useful for the prediction and early detection of disorders in mothers and babies.
* Analyze infant neurodevelopment and psychopathology during the first two years of life.

METHODOLOGY:

1. Design: A randomized clinical trial, blinded to the investigator, with two parallel groups (1 experimental group using the digital tool and 1 control group).

   The protocol has been designed following the CONsolidated Standards Of Reporting Trials (CONSORT: http://www.consortstatement.org) and the Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT).
2. Participants: The study will be conducted at Vall d'Hebrón Hospital, the Sexual and Reproductive Health Care Services (ASSIR) in Tarragona, ASSIR del Litoral (Barcelona), and Hospital del Mar.

   Participants will be pregnant women between 12-14 weeks of gestation who are following their pregnancy at these centers, and they and their babies will be followed up until 24 months postpartum.
3. Sample Size: To estimate the necessary sample size to detect significant differences between groups, an alpha risk error of 0.05 and a beta risk error of 0.2 for one-tailed tests have been accepted, considering a dropout rate of 40%. According to data from Viskovich et al. (2020) and Rash et al. (2011) related to the Satisfaction With Life Scale, 16 subjects per group are needed to determine minimum differences of 1.86 points, assuming a standard deviation of 2.07 points. According to data from Tovote et al. (2014) related to the World Health Organization-5 Well-Being Index, 11 subjects per group are needed to determine minimum differences of 20.6 points, assuming a standard deviation of 19.0 points. According to data from Ahlqvist-Björkroth et al. (2019) related to the Edinburgh Postnatal Depression Scale, 26 subjects per group are needed to determine minimum differences of 2.13 points, assuming a standard deviation of 2.46 points. Finally, according to data from Moix et al. (2021) related to the State-Trait Anxiety Inventory, 11 subjects per group are needed to determine minimum differences of 5.54 points, assuming a standard deviation of 4.5 points. Thus, 64 subjects per arm are needed, so a total sample of 300 pregnant women per center should be recruited.
4. Procedures:

4.1. Recruitment: Participants will be recruited through midwives from the Primary Care Centers and Sexual and Reproductive Health Care Services (ASSIR) of Tarragona, and ASSIR of Barcelona Litoral - Hospital del Mar. Recruitment will be through obstetricians and midwives from the same center. Women who visit before 15 weeks of gestation and meet the inclusion and exclusion criteria will be eligible to participate in the study. The healthcare professional conducting the visit will be responsible for validating the inclusion and exclusion criteria.

4.2. Randomization: Balanced randomization by center will be carried out through the digital tool itself, so the researchers will be blind to the intervention. Participants will need to download the mobile application, where during the registration process and center selection, they will be randomized into the control or intervention group. Women in the intervention group will be offered access to the full digital tool, while those in the control group will have an app with no content.

4.3. Blinding: Researchers analyzing the primary data and conducting infant evaluations will not know which group the women have been assigned to. Midwives and obstetricians who conduct recruitment will also be unaware, unless the participant discloses it after being randomized. Neither the researchers nor the midwives will have access to group assignments. Researchers conducting primary data analysis or neonatal evaluations will not know the participants' group assignments until the end of the study. Due to the nature of the intervention, participants cannot be blinded to their group assignment.

4.4. Pseudonymization: Data pseudonymization and protection will be ensured using the REDCap system. Each participating health center and hospital (as independent data controllers) will have access only to their own center's data, not to data from other centers. Data from the entire study recorded in REDCap and app data will be accessible only by the co-sponsors and co-controllers of the data mentioned in the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 12-14 weeks of gestation.
* The first obstetric ultrasound has been performed.
* Women who know how to read and understand Spanish.
* Women who have access to a mobile phone with an internet connection (data or wifi)
* Women who have knowledge of technology tools via app.
* Have signed the informed consent to participate in the study.

Exclusion Criteria:

* Termination of pregnancy, or early miscarriage
* Perinatal loss at any time during pregnancy.
* Severe mental pathology or moderate unstable mental pathology.
* Consumption of toxic substances.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnancy
Enrollment: 1200 (Estimated)
Dates: Start 2024-12-28 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Maternal well-being | 12-14 weeks, 33-34 weeks of gestation, 6 weeks, 6, 12, 24 months postpartum.
  Assessed using the World Health Organization-5 Well-Being Index (WHO-5). The WHO-5 is a brief 5-item self-report instrument designed to measure current mental well-being. It has adequate validity for screening depression and measuring clinical trial outcomes, with good properties when used in pregnant women (Mortazavi et al., 2021).
  Min value: 0 Max value: 25 Higher scores: Indicate better well-being. Scores below 13 suggest poor well-being, indicative of depression.

SECONDARY OUTCOMES:
Depression | 12-14 and 29-30 weeks of pregnancy, 6 weeks, 6, 12, 24 months postpartum.
  Using the Edinburgh Postpartum Depression Scale (EPDS), a 10-item questionnaire for detecting postpartum depression symptoms, validated for pregnancy and in Spanish women (Levis et al., 2020; Vázquez & Míguez, 2019).
  Min value: 0 Max value: 30 Higher scores: Indicate worse symptoms. Scores ≥10 suggest possible depression; scores ≥13 or positive for question 10 indicate a high likelihood.
Anxiety | 12-14 and 33-34 weeks of pregnancy, 6 weeks, 6, 12, 24 months postpartum.
  Using the State-Trait Anxiety Inventory (STAI), a 40-item tool for assessing state and trait anxiety (Brunton et al., 2015).
  Min value: 20 per subscale (STAI-S and STAI-T) Max value: 80 per subscale Higher scores: Indicate worse anxiety outcomes.
Birth Fear | 12-14 and 33-34 weeks of pregnancy, 6 weeks postpartum.
  Using the Wijma Delivery Expectancy/Experience Questionnaire (W-DEQ A-B), a 33-item tool to quantify fear of childbirth.
  Min value: 0 Max value: 165 Higher scores: Indicate higher levels of fear; scores >85 suggest high fear levels.
Sleep | 12-14 and 33-34 weeks of pregnancy
  Using the Pittsburgh Sleep Quality Index (PSQI), a 19-item tool to assess sleep quality over the past 30 days.
  Min value: 0 Max value: 21 Higher scores: Indicate worse sleep quality; scores >5 suggest poor sleep.
Maternal Antenatal attachment | 29-30 weeks of pregnancy.
  Using the Maternal Antenatal Attachment Scale (MAAS) to assess the emotional bond with the unborn child.
  Min value: 19 Max value: 95 Higher scores: Indicate a stronger emotional bond.
Bonding | 6 weeks, 6, 12, 24 months postpartum.
  Using the Postpartum Bonding Questionnaire (PBQ) to measure the maternal bond with the baby post-birth.
  Min value: 0 Max value: 125 Higher scores: Indicate worse bonding outcomes.
Birth Experience | 33-34 weeks of pregnancy, 6 weeks postpartum.
  Using the Mackey Satisfaction Childbirth Questionnaire to measure childbirth satisfaction.
  Min value: 11 Max value: 55 Higher scores: Indicate higher satisfaction.
Traumatic stress responses related to childbirth | 6 weeks postpartum
  The City Birth Trauma Scale (BiTS): Psychological assessment tool designed to measure traumatic stress responses specifically related to childbirth. It is used to identify symptoms of birth-related post-traumatic stress disorder (PTSD) in women who have recently given birth. The scale helps healthcare providers to assess the severity and impact of traumatic childbirth experiences on mothers.
  Minimum value: 0 Maximum value: 80 Higher scores: Indicate more severe symptoms of trauma related to childbirth.
Parental stress | 6, 12, 24 months postpartum.
  Parental Stress Index (PSI): This evaluation tool measures parental stress levels in mothers and fathers. The PSI consists of 36 questions that evaluate different factors that may contribute to parental stress, such as the child's health, the relationship with the partner, social support, work demands, and parental expectations regarding the child's development.
  Min value: 36 Max value: 180 Higher scores: Indicate higher stress levels.
Maternal empowerment | Postpartum: 6 weeks and 24 months
  Parenting Sense of Competence (PSOC): This evaluation tool measures the perception of parental competence in mothers and fathers. The PSOC consists of 16 questions that evaluate satisfaction with the parental role, confidence in parenting skills, the ability to adapt to the child's demands, and the perception that the parental role is a rewarding task. The questionnaire is used to identify parents who may need additional support to develop confidence and parenting skills, and improve family health and well-being.
  Minimum value: 16 Maximum value: 96 Higher scores: Indicate better perceived parental competence.
Physical Activity | 12-14 and 33-34 weeks of pregnancy.
  Using the International Physical Activity Questionnaire (IPAQ) to measure physical activity levels.
  Min value: 0 Max value: Varies based on intensity and frequency Higher scores: Indicate higher physical activity levels.
Pregnancy outcomes | 1 week after birth collected retrospectively for pregnancy and childbirth
  Pregnancy complications (measured in presence of gestational diabetes, preeclampsia, preterm birth, growth restriction, diagnosis of perinatal mental health disorder, need for psychotropic drugs, smoking habit).
  Higher values: Indicate higher complications during pregnancy.
Health costs 1 | 1 week after birth collected retrospectively for pregnancy and childbirth. 2 years postnatally collected retrospectively for the postnatal period.
  Cost for the healthcare system (measured on number of visits to obstetrician/gynecology, midwife, psychology, physiotherapy, emergency room, hospital admissions)
  Higher values: Indicate higher expenses for the healthcare system.
Health costs 2 | 1 week after birth collected retrospectively for pregnancy and childbirth. 2 years postnatally collected retrospectively for the postnatal period.
  Duration of hospital admission (measured in days).
  Higher values: Indicate higher expenses for the healthcare system.
Neonatal outcomes 1 | 1 week after birth collected retrospectively
  Gestational age at delivery (weeks+days) Normal range: 37-42 weeks Lower values: Indicate preterm newborns. Higher values: Indicate postterm newborns.
Neonatal outcomes 2 | 1 week after birth collected retrospectively
  Cord arterial pH (potential of hydrogen)
  Normal pH:
  Range: 7.25 to 7.35 Implication: Indicates that the newborn had adequate oxygenation and no significant acidosis during labor and delivery.
  Mild Acidosis:
  Range: 7.20 to 7.24 Implication: Suggests a slight decrease in oxygen levels. While it may not immediately be cause for concern, it warrants monitoring for any signs of distress or complications.
  Moderate Acidosis:
  Range: 7.10 to 7.19 Implication: Indicates moderate hypoxia and the possibility of metabolic acidosis. This condition may require intervention and close monitoring of the newborn for any further complications.
  Severe Acidosis:
  Range: Below 7.10 Implication: Suggests significant hypoxia and severe metabolic acidosis, which can be associated with perinatal asphyxia. Immediate medical evaluation and intervention are typically required to address any potential adverse outcomes.
Neonatal outcomes 3 | 1 week after birth collected retrospectively
  Neonatal complications at birth (descriptive: admission to the ICU, neonatal sepsis)
Neonatal outcomes 4 | 1 week after birth collected retrospectively
  Apgar score: The Apgar score is a quick test performed on a newborn at 1 minute and 5 minutes after birth. The purpose of the test is to determine how well the baby tolerated the birthing process and how well the baby is doing outside the mother's womb.
  The Apgar score assesses five criteria, each scored on a scale of 0 to 2, with a maximum total score of 10:
  Score 7-10: Generally considered normal; indicates that the newborn is in good health.
  Score 4-6: Fairly low; may require some medical intervention such as oxygen or physical stimulation.
  Score 0-3: Critically low; requires immediate resuscitation and medical attention.
Neonatal outcomes 5 | 1 week after birth collected retrospectively
  Weight (in grams)
Neonatal outcomes 6 | 1 week after birth collected retrospectively
  Height (centimeters)
Neonatal outcomes 7 | 1 week after birth collected retrospectively
  Head circumference (centimeters)
Birth outcomes 1 | 1 week after birth collected retrospectively
  Type of birth. Measures in normal vaginal birth, instrumental birth and caesarian section.
Birth outcomes 2 | 1 week after birth collected retrospectively
  State of the perineum after delivery: Measured in intact perineum, I degree tear, II degree tear, III degree tear, IV degree tear and episiotomy.
Birth outcomes 3 | 1 week after birth collected retrospectively
  Type of analgesia during delivery: measured in epidural (yes/no), raquideal (yes/no), local (yes/no), and general (yes/no)
Birth outcomes 4 | 1 week after birth collected retrospectively
  Labor induction: Descriptive yes/no
Birth outcomes 5 | 1 week after birth collected retrospectively
  Maternal complications at birth (descriptive: admission to the ICU, obstetric emergency)
Biomarkers 1 (stress) | From 12 weeks of pregnancy until 2 years postpartum
  Maternal heart rate variability (HRV)
  Heart rate:
  Minimum Value: Varies depending on the individual's baseline, but generally, a healthy resting heart rate for adults ranges from 60 to 100 beats per minute (bpm).
  Maximum Value: This can vary widely based on activity and stress levels, but for pregnant women, a heart rate consistently above 100 bpm at rest might be concerning
  Maternal heart rate variability (HRV) refers to the variation in time intervals between heartbeats, which is a marker of autonomic nervous system function.
  Minimum Value: HRV does not have a fixed minimum value, but lower HRV generally indicates reduced autonomic flexibility and poor cardiovascular health.
  Maximum Value: Similarly, there is no fixed maximum value, but higher HRV is generally associated with better cardiovascular fitness and autonomic regulation.
Biomarkers 2 (sleep) | From 12 weeks of pregnancy until 2 years postpartum
  Sleeping patterns (measured with wearable):
  Key Metrics Monitored by Wearable:
  Sleeping patterns refer to the habitual sleep behaviors of an individual. Bed time start (date and time), bed time end (date and time) and awake time (in minutes) will be combined to report total sleep (in minutes).
  The overall of this metrics will give a score for sleeping patterns. Higher levels mean higher levels of resting.
Biomarkers 3 (activity) | From 12 weeks of pregnancy until 2 years postpartum
  Level of physical activity (measured with wearable):
  The heart rate monitor of the wearable measures the wearer's heart rate to gauge intensity of physical activity.
  The amount of time (in minutes) will give us the time a day spent in physical activities of moderate or higher intensity (HR>100bpm).
  Higher levels mean higher levels of physical activity.
Child neurodevelopment | 6 months, 12 months and 24 months postpartum.
  Ages and Stages Questionnaires (ASQ): This evaluation tool measures child development in areas such as communication, social behavior, motor coordination, language, and learning. The ASQ consists of different questionnaires adapted to different ages, which are completed by parents or caregivers. The results are used to identify children with potential developmental delays and provide early interventions to improve their cognitive and emotional health. The ASQ is widely used in clinical practice and research in the field of child development.
  Scores vary across different developmental domains: Communication, Social Behavior, Motor Coordination, Language, Learning.
  Higher scores: Indicate better developmental outcomes .
Child neurodevelopment | 4 months and 24 months postpartum.
  The Bayley Scales of Infant and Toddler Development, commonly referred to as the Bayley Scales, is a standardized assessment tool used to evaluate the developmental functioning of infants and toddlers, typically from 1 month to 42 months of age.
  The Bayley Scales consist of five key domains, each designed to measure different aspects of a child's development: cognitive, language, motor, social-emotional and adaptive behaviour.
  The result is presented in percentiles (0-100)
  Higher scores: Indicate better developmental outcomes.
Adaptative behaviour | 4 months and 24 months postpartum.
  Vineland III: This evaluation tool is designed to measure adaptive skills in individuals of all ages, from infancy to adulthood.
  Scores vary across different subscales: Communication Skills, Social Skills, Daily Living Skills.
  Higher scores: Indicate better adaptive functioning.
Breastfeeding outcomes | 1 week after birth collected retrospectively
  Type of breastfeeding at discharge from hospital. Descriptive outcome reported as exclusive breastfeeding, mixed feeding or artificial feeding.
Breastfeeding outcomes | Postpartum: 4 months, 1 year after childbirth collected retrospectively
  Breastfeeding duration (measured in days)

CONTACTS AND LOCATIONS:
Overall Officials: Roser Palau-Costafreda, PhD, Principal Investigator — A Thousand Colibris, S.L
Locations (3):
- Spain (3):
  - Hospital Vall d'Hebron, Barcelona, Catalonia
  - Hospital del Mar, Barcelona
  - ASSIR Tarragona, Tarragona

IPD SHARING:
Plan to Share IPD: No
The data-sharing plans for the current study are unknown and will be made available at a later date.

REFERENCES:
- [Background] Uguz F, Yakut E, Aydogan S, Bayman MG, Gezginc K. Prevalence of mood and anxiety disorders during pregnancy: A case-control study with a large sample size. Psychiatry Res. 2019 Feb;272:316-318. doi: 10.1016/j.psychres.2018.12.129. Epub 2018 Dec 25. PMID 30597383
- [Background] Glover, V., Ahmed-Salim, Y., &amp;amp;amp;amp;amp; Capron, L. (2016). Maternal anxiety, depression, and stress during pregnancy: Effects on the fetus and the child, and underlying mechanisms. In Fetal Development: Research on Brain and Behavior, Environmental Influences, and Emerging Technologies (pp. 213-227). Springer International Publishing. https://doi.org/10.1007/978-3-319-22023-9_12
- [Background] Glover V. Effects of Maternal Prenatal Stress on the Fetal Brain and Hope for the Prevention of Psychopathology. Biol Psychiatry. 2020 Mar 15;87(6):487-488. doi: 10.1016/j.biopsych.2019.11.008. No abstract available. PMID 32081251
- [Background] Fairbrother N, Young AH, Janssen P, Antony MM, Tucker E. Depression and anxiety during the perinatal period. BMC Psychiatry. 2015 Aug 25;15:206. doi: 10.1186/s12888-015-0526-6. PMID 26303960
- [Background] Evans K, Morrell CJ, Spiby H. Systematic review and meta-analysis of non-pharmacological interventions to reduce the symptoms of mild to moderate anxiety in pregnant women. J Adv Nurs. 2018 Feb;74(2):289-309. doi: 10.1111/jan.13456. Epub 2017 Oct 16. PMID 28921612
- [Background] Cena L, Gigantesco A, Mirabella F, Palumbo G, Trainini A, Stefana A. Prevalence of Maternal Postnatal Anxiety and Its Association With Demographic and Socioeconomic Factors: A Multicentre Study in Italy. Front Psychiatry. 2021 Sep 30;12:737666. doi: 10.3389/fpsyt.2021.737666. eCollection 2021. PMID 34658970
- [Background] Beddoe AE, Lee KA. Mind-body interventions during pregnancy. J Obstet Gynecol Neonatal Nurs. 2008 Mar-Apr;37(2):165-75. doi: 10.1111/j.1552-6909.2008.00218.x. PMID 18336440
- [Background] Alder J, Fink N, Bitzer J, Hosli I, Holzgreve W. Depression and anxiety during pregnancy: a risk factor for obstetric, fetal and neonatal outcome? A critical review of the literature. J Matern Fetal Neonatal Med. 2007 Mar;20(3):189-209. doi: 10.1080/14767050701209560. PMID 17437220
- [Background] Yuen WS, Lo HC, Wong WN, Ngai FW. The effectiveness of psychoeducation interventions on prenatal attachment: A systematic review. Midwifery. 2022 Jan;104:103184. doi: 10.1016/j.midw.2021.103184. Epub 2021 Oct 28. PMID 34753018
- [Background] Woody CA, Ferrari AJ, Siskind DJ, Whiteford HA, Harris MG. A systematic review and meta-regression of the prevalence and incidence of perinatal depression. J Affect Disord. 2017 Sep;219:86-92. doi: 10.1016/j.jad.2017.05.003. Epub 2017 May 8. PMID 28531848
- [Background] Veringa IK, de Bruin EI, Bardacke N, Duncan LG, van Steensel FJ, Dirksen CD, Bogels SM. 'I've Changed My Mind', Mindfulness-Based Childbirth and Parenting (MBCP) for pregnant women with a high level of fear of childbirth and their partners: study protocol of the quasi-experimental controlled trial. BMC Psychiatry. 2016 Nov 7;16(1):377. doi: 10.1186/s12888-016-1070-8. PMID 27821151
- [Background] Van den Bergh BRH, van den Heuvel MI, Lahti M, Braeken M, de Rooij SR, Entringer S, Hoyer D, Roseboom T, Raikkonen K, King S, Schwab M. Prenatal developmental origins of behavior and mental health: The influence of maternal stress in pregnancy. Neurosci Biobehav Rev. 2020 Oct;117:26-64. doi: 10.1016/j.neubiorev.2017.07.003. Epub 2017 Jul 28. PMID 28757456
- [Background] van Agteren J, Iasiello M, Lo L, Bartholomaeus J, Kopsaftis Z, Carey M, Kyrios M. A systematic review and meta-analysis of psychological interventions to improve mental wellbeing. Nat Hum Behav. 2021 May;5(5):631-652. doi: 10.1038/s41562-021-01093-w. Epub 2021 Apr 19. PMID 33875837
- [Background] Urech C, Fink NS, Hoesli I, Wilhelm FH, Bitzer J, Alder J. Effects of relaxation on psychobiological wellbeing during pregnancy: a randomized controlled trial. Psychoneuroendocrinology. 2010 Oct;35(9):1348-55. doi: 10.1016/j.psyneuen.2010.03.008. Epub 2010 Apr 22. PMID 20417038
- [Background] Steptoe A, Deaton A, Stone AA. Subjective wellbeing, health, and ageing. Lancet. 2015 Feb 14;385(9968):640-648. doi: 10.1016/S0140-6736(13)61489-0. Epub 2014 Nov 6. PMID 25468152
- [Background] Stein A, Pearson RM, Goodman SH, Rapa E, Rahman A, McCallum M, Howard LM, Pariante CM. Effects of perinatal mental disorders on the fetus and child. Lancet. 2014 Nov 15;384(9956):1800-19. doi: 10.1016/S0140-6736(14)61277-0. Epub 2014 Nov 14. PMID 25455250
- [Background] Smith A, Twynstra J, Seabrook JA. Antenatal depression and offspring health outcomes. Obstet Med. 2020 Jun;13(2):55-61. doi: 10.1177/1753495X19843015. Epub 2019 Apr 24. PMID 32714436
- [Background] Sadler LS, Slade A, Close N, Webb DL, Simpson T, Fennie K, Mayes LC. Minding the Baby: Enhancing reflectiveness to improve early health and relationship outcomes in an interdisciplinary home visiting program. Infant Ment Health J. 2013 Sep 1;34(5):391-405. doi: 10.1002/imhj.21406. PMID 24049219
- [Background] Pearson RM, Carnegie RE, Cree C, Rollings C, Rena-Jones L, Evans J, Stein A, Tilling K, Lewcock M, Lawlor DA. Prevalence of Prenatal Depression Symptoms Among 2 Generations of Pregnant Mothers: The Avon Longitudinal Study of Parents and Children. JAMA Netw Open. 2018 Jul 6;1(3):e180725. doi: 10.1001/jamanetworkopen.2018.0725. PMID 30646025
- [Background] Oyarzabal EA, Seuferling B, Babbar S, Lawton-O'Boyle S, Babbar S. Mind-Body Techniques in Pregnancy and Postpartum. Clin Obstet Gynecol. 2021 Sep 1;64(3):683-703. doi: 10.1097/GRF.0000000000000641. PMID 34162789
- [Background] Muller M, Matthies LM, Goetz M, Abele H, Brucker SY, Bauer A, Graf J, Zipfel S, Hasemann L, Wallwiener M, Wallwiener S. Effectiveness and cost-effectiveness of an electronic mindfulness-based intervention (eMBI) on maternal mental health during pregnancy: the mindmom study protocol for a randomized controlled clinical trial. Trials. 2020 Nov 17;21(1):933. doi: 10.1186/s13063-020-04873-3. PMID 33203471
- [Background] Morres ID, Tzouma NA, Hatzigeorgiadis A, Krommidas C, Kotronis KV, Dafopoulos K, Theodorakis Y, Comoutos N. Exercise for perinatal depressive symptoms: A systematic review and meta-analysis of randomized controlled trials in perinatal health services. J Affect Disord. 2022 Feb 1;298(Pt A):26-42. doi: 10.1016/j.jad.2021.10.124. Epub 2021 Oct 30. PMID 34728280
- [Background] Khoury B, Lecomte T, Fortin G, Masse M, Therien P, Bouchard V, Chapleau MA, Paquin K, Hofmann SG. Mindfulness-based therapy: a comprehensive meta-analysis. Clin Psychol Rev. 2013 Aug;33(6):763-71. doi: 10.1016/j.cpr.2013.05.005. Epub 2013 Jun 7. PMID 23796855
- [Background] Huguet A, Rao S, McGrath PJ, Wozney L, Wheaton M, Conrod J, Rozario S. A Systematic Review of Cognitive Behavioral Therapy and Behavioral Activation Apps for Depression. PLoS One. 2016 May 2;11(5):e0154248. doi: 10.1371/journal.pone.0154248. eCollection 2016. PMID 27135410
- [Background] Hernandez-Martinez C, Val VA, Murphy M, Busquets PC, Sans JC. Relation between positive and negative maternal emotional states and obstetrical outcomes. Women Health. 2011 Mar;51(2):124-35. doi: 10.1080/03630242.2010.550991. PMID 21476173
- [Background] Hernandez-Martinez C, Arija V, Balaguer A, Cavalle P, Canals J. Do the emotional states of pregnant women affect neonatal behaviour? Early Hum Dev. 2008 Nov;84(11):745-50. doi: 10.1016/j.earlhumdev.2008.05.002. Epub 2008 Jun 20. PMID 18571345
- [Background] Goodman JH, Guarino A, Chenausky K, Klein L, Prager J, Petersen R, Forget A, Freeman M. CALM Pregnancy: results of a pilot study of mindfulness-based cognitive therapy for perinatal anxiety. Arch Womens Ment Health. 2014 Oct;17(5):373-87. doi: 10.1007/s00737-013-0402-7. Epub 2014 Jan 22. PMID 24449191
- [Background] Goodman JH, Chenausky KL, Freeman MP. Anxiety disorders during pregnancy: a systematic review. J Clin Psychiatry. 2014 Oct;75(10):e1153-84. doi: 10.4088/JCP.14r09035. PMID 25373126
- [Background] Firth J, Torous J, Nicholas J, Carney R, Pratap A, Rosenbaum S, Sarris J. The efficacy of smartphone-based mental health interventions for depressive symptoms: a meta-analysis of randomized controlled trials. World Psychiatry. 2017 Oct;16(3):287-298. doi: 10.1002/wps.20472. PMID 28941113
- [Background] Espie CA, Emsley R, Kyle SD, Gordon C, Drake CL, Siriwardena AN, Cape J, Ong JC, Sheaves B, Foster R, Freeman D, Costa-Font J, Marsden A, Luik AI. Effect of Digital Cognitive Behavioral Therapy for Insomnia on Health, Psychological Well-being, and Sleep-Related Quality of Life: A Randomized Clinical Trial. JAMA Psychiatry. 2019 Jan 1;76(1):21-30. doi: 10.1001/jamapsychiatry.2018.2745. PMID 30264137
- [Background] Domhardt M, Gesslein H, von Rezori RE, Baumeister H. Internet- and mobile-based interventions for anxiety disorders: A meta-analytic review of intervention components. Depress Anxiety. 2019 Mar;36(3):213-224. doi: 10.1002/da.22860. Epub 2018 Nov 19. PMID 30450811
- [Background] Closa-Monasterolo R, Gispert-Llaurado M, Canals J, Luque V, Zaragoza-Jordana M, Koletzko B, Grote V, Weber M, Gruszfeld D, Szott K, Verduci E, ReDionigi A, Hoyos J, Brasselle G, Escribano Subias J. The Effect of Postpartum Depression and Current Mental Health Problems of the Mother on Child Behaviour at Eight Years. Matern Child Health J. 2017 Jul;21(7):1563-1572. doi: 10.1007/s10995-017-2288-x. PMID 28188472
- [Background] Chung KF, Lee CT, Yeung WF, Chan MS, Chung EW, Lin WL. Sleep hygiene education as a treatment of insomnia: a systematic review and meta-analysis. Fam Pract. 2018 Jul 23;35(4):365-375. doi: 10.1093/fampra/cmx122. PMID 29194467
- [Background] Battulga B, Benjamin MR, Chen H, Bat-Enkh E. The Impact of Social Support and Pregnancy on Subjective Well-Being: A Systematic Review. Front Psychol. 2021 Sep 9;12:710858. doi: 10.3389/fpsyg.2021.710858. eCollection 2021. PMID 34566789
- [Background] Arranz Freijo, E., Olabarrieta, F., Manzano, A., Barreto, F. B., Roncallo, C. P., Sánchez Murciano, M., Rekagorri, J., &amp;amp;amp;amp;amp;amp;amp;amp;amp;amp;amp; Garcia, M. D. (2019). Assessment and preventive education for families, based on the principles of positive parenting. Early Child Development and Care, 189(5), 792-801. https://doi.org/10.1080/03004430.2017.1344234
- See also: Study Website: MamaConecta is the name under which we publicly present the clinical study investigating perinatal mental health and the impact of digital health tools on prevention and treatment. The co-promoters of this study are A THOUSAND COLIBRIS S.L — https://mamaconecta.com/